CLINICAL TRIAL: NCT03393650
Title: Effect of Protein Supplementation Combined With Mixed Power Training on Muscle Function, Composition, Phenotype and Functional Capacities Compared to Mixed Power Training Alone in Elderly Men
Brief Title: Protein Supplementation and Mixed Power Training on Muscle Function and Functional Capacities in Elderly Men
Acronym: PROMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Responsible Party: Principal Investigator, Mylène Aubertin-Leheudre, Professor, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UQAM
Record Dates: First submitted 2016-12-15; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Dynapenia; Aging; Physical Impairment
Keywords: exercise; protein; muscle function; aging
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise + Placebo group (Active Comparator): 50 subjects will receive a placebo supplementation with an exercise intervention (EX group)
  Interventions: Other: Exercise + Placebo group
- Exercise + Protein group (Active Comparator): 50 subjects will receive a protein supplementation combined with an exercise intervention (PROTEX group)
  Interventions: Other: Exercise + Protein group

INTERVENTIONS:
Other: Exercise + Placebo group — 1/2 of the subject will follow a mixed power training: 4 power exercises + 6 functional exercises combined to a placebo
  Arms: Exercise + Placebo group
Other: Exercise + Protein group — 1/2 of the subject will receive 30 g/ d of protein (leucine+ vitD; divided in three equal doses: morning, afternoon and evening) + will follow a mixed power training: 4 power exercises + 6 functional exercises.
  Arms: Exercise + Protein group

SUMMARY:
Investigate the effect of 12 weeks mixed power training (power and functional exercises) combined with a protein supplementation (30g/d) or not (placebo) on physiological characteristics of muscle and functional capacities in elderly men.

DETAILED DESCRIPTION:
Life habits are know to be able to prevent the loss of functional capacities and muscle function during aging process. More specifically, protein intake is important to maintain muscle function in older adults. Another non pharmacological intervention and well recognized for its efficacy, it's exercise training.

Recently, it has been observed than muscle quality is more important to maintain physical autonomy than muscle mass per se. In addition, muscle quality is more related to functional capacities than muscle mass.

Due to this recent finding, it has been proposed that muscle power training would be the best exercise intervention to prevent the loss of mobility.

ELIGIBILITY:
Inclusion Criteria:

* Elderly men
* 60 years and older
* Sedentary men
* Not obese (BMI <30 kg/m2)
* Living in free-living community

Exclusion Criteria:

* Not able to follow an exercise program (doctor authorization: XAAP)
* Having Lactose intolerance
* Having Pace marker
* Having Metabolism disorder
* No weight stable since the last 6 months
* No stable medication (same dose and type since at least 6 months)

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in walking speed | Change from Baseline walking speed at 12 weeks measure in all subjects
  evaluate using the 4m- normal walking speed (m/sec)

SECONDARY OUTCOMES:
Change in lower limb muscle quality | Change from Baseline lower limb muscle quality at 12 weeks measure in all subjects
  Knee extension muscle strength (isometric (N)/ lower limb muscle mass (kg))

OTHER OUTCOMES:
Change in mitochondrial activity | Change from Baseline mitochondrial activity at 12 weeks measure in half of the subjects
  citrate synthase activity (unit: percent)

CONTACTS AND LOCATIONS:
Overall Officials: mylene aubertin-leheudre, PhD, Principal Investigator — Université du Québec a Montréal

IPD SHARING:
Plan to Share IPD: Undecided